CLINICAL TRIAL: NCT05021913
Title: A Clinical Study to Evaluate the Safety and Performance of DKL Crosslinked Sodium Hyaluronate 23 Dermal Filler for Improvement of Nasolabial Fold Appearance
Brief Title: Safety and Performance of DKL Crosslinked Sodium Hyaluronate 23 Dermal Filler for Improvement of NLF Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Korman Laboratories Ltd. (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAL-P68
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Aging, Premature
Keywords: Premature skin aging; Correction of facial structural defects; Wrinkles
MeSH Terms: conditions — Aging, Premature

STUDY DESIGN:
Intervention Model Description: Pivotal, prospective, active-controlled, randomized, double blinded (blinded evaluator and subject), intra-individual split-face comparison
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double blinded (blinded evaluator and subject) study and the allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device (Experimental): DKL crosslinked sodium hyaluronate 23
  Interventions: Device: DKL crosslinked sodium hyaluronate 23
- Comparator product (Active Comparator): Juvéderm Volift™ with lidocaine (Allergan, Inc)
  Interventions: Device: Juvéderm Volift™ with lidocaine (Allergan, Inc)

INTERVENTIONS:
Device: DKL crosslinked sodium hyaluronate 23 — is injected into the NLF on Day 1. The volume of injection will not exceed 2 mL per side. If applicable, a touch-up of DKL crosslinked sodium hyaluronate 23 will be injected on Day 30; the volume of injection will not exceed 1 mL per side.
  Arms: Investigational device
Device: Juvéderm Volift™ with lidocaine (Allergan, Inc) — is injected into the NLF on Day 1. The volume of injection will not exceed 2 mL per side. If applicable, a touch-up of Juvéderm Volift™ will be injected on Day 30; the volume of injection will not exceed 1 mL per side.
  Arms: Comparator product

SUMMARY:
This is a pivotal, prospective active-controlled, randomized, double blinded (blinded evaluator and subject), intra-individual split-face comparison, non-inferiority study of DKL crosslinked sodium hyaluronate 23 versus Juvederm Volift™ after injection into the mid to deep dermis for correction of moderate to deep nasolabial folds (NLFs).

DETAILED DESCRIPTION:
This is a pivotal, prospective active-controlled, randomized, double blinded (blinded evaluator and subject), intra-individual split-face comparison, non- inferiority study of DKL crosslinked sodium hyaluronate 23 versus Juvederm Volift™ after injection into the mid to deep dermis for correction of moderate to deep nasolabial folds (NLFs).

Approximately 40 subjects will be randomized and treated. Subjects will come to the research clinic for up to 6 visits, including a screening/baseline visit and up to 5 follow-up visits.

At Screening eligible subjects (males and females aged 18 to 65 years) will be randomized as to which NLF will be treated with the investigational device and which NLF will be treated with the comparator device.

The subjects will undergo baseline assessments of NLF Wrinkle Severity Rating Scale (WSRS) by the evaluating investigator and have baseline two-dimensional (2D) photos taken, prior to treatment with the investigational device and comparator.

Treatment will be performed by an unblinded treating investigator. Following treatment, the subjects will complete a subject eDiary in which they will assess pre-defined treatment related events experienced during the first 14 days after the injection.

Additional visits will take place 1, 3, 6 and 9 months after the treatment. During these visits the subjects will undergo evaluations by an evaluating investigator blinded to the treatment allocation. Assessments will include photography, NLF WSRS and Global Aesthetic Improvement Scale (GAIS). The subjects will also evaluate treatment outcome using the GAIS and complete a patient satisfaction questionnaire. The investigator will record any adverse events (AEs) that have occurred and will note their severity and relationship to the injected product.

An optional touch-up treatment will be performed one month after the initial treatment at the discretion of the treating investigator. Subjects requiring touch-up will receive touch-up according to the original randomization scheme, i.e. the investigational device and comparator product will be injected to the same NLF according to the randomization scheme. Following touch-up, these subjects will be asked to complete a subject eDiary for assessment of pre-defined treatment related events experienced during the first 14 days after the injection. Subjects receiving touch-up will attend and additional evaluation visit one month after touch-up (in addition to other visits).

The treating investigators will complete a usability questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Review and sign the Independent Ethics Committee (IEC)-approved Informed Consent Form (ICF) prior to any study-related procedures being performed. In addition, the subject will be asked to provide a separate release for use of their photographs in publications and the clinical investigation report (CIR). The subject has a right to refuse the photo release without jeopardizing their eligibility to participate in the study.
2. Male and female subjects aged 18 to 65 years (inclusive) at the time of screening.
3. Subject desires correction of NLFs.
4. Moderate to severe bilateral aging defects in the nasolabial area, with wrinkles classified as grade 3 or 4 according to the NLF WSRS on each side as assessed by the blinded evaluator. NLFs should be of the same grade on the left and right side of the face (i.e. approximate bilateral symmetry).
5. Subject, that in the opinion of the blinded evaluator, can improve at least 1 step on the investigator-rated NLF WSRS with a maximum volume of 2.0 mL/NLF for initial treatment and 1.0 mL/NLF for touch-up.
6. Female of child-bearing potential (sexually active and not sterile nor postmenopausal for at least 1 year) should have a urine pregnancy test evaluated as negative on the day of enrolment, and agree to use a reliable method of contraception for the duration of the study (effective birth control measures include sexual abstinence, combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS] and/or condom with spermicide).
7. Subject agrees to abstain from any facial cosmetic or surgical procedures during the study period.
8. Subject agrees to refrain from excessive weight gain or loss (±10%) during the investigation period.
9. Subject has adequate understanding of the local language to understand verbal and written subject information and is willing to comply with the study requirements.

Exclusion Criteria:

1. History of any clinically significant disease or disorder, including porphyria or systemic disorders affecting wound healing, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational device and comparator.
3. History of anaphylaxis, multiple severe allergies, atopy, or allergy to sodium hyaluronate products or to streptococcal proteins or have plans to undergo desensitization therapy during the term of the study.
4. History of immune system disorders (e.g., autoimmune disease, human immunodeficiency virus [HIV]-positive status, history of immune system degradation, or recurrent herpes simplex).
5. History of streptococcal disease (e.g. recurrent sore throat) and subjects with rheumatic fever, as judged by the investigator.
6. Dermatological problems (e.g. cutaneous lesions, inflammatory skin conditions, hypertrophic scars or a tendency for keloid formation) at the discretion of the investigator.
7. Noticeable scarring (including acne scarring), prior surgery, an active inflammation, infection, cancerous or pre-cancerous lesion, history of prior significant trauma to the midface, such as dog bite or laceration, resulting in formation of a scar, or unhealed wound or have undergone radiation treatment in the area to be treated.
8. Cheek tattoos, piercings, facial hair, or scars that would interfere with visualization of the cheek area for the effectiveness assessments.
9. Very thin skin in the mid-facial region, tendency to accumulate fluid in the lower eyelids, or large infraorbital fat pads, i.e., significant convexity or projection from the infraorbital fat pads.
10. Mid-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease or HIV-related disease.
11. Moderate or severe abnormal midface or cheek asymmetry.
12. Ongoing or history of use of immunosuppressive therapy.
13. Use of anti-coagulation, anti-platelet, or thrombolytic medications, anti-inflammatory drugs, or other substances known to increase coagulation time (as detailed in Section 9.6.2) within 10 days prior to treatment with the investigational device and comparator.
14. Use of any new (i.e. that the subject has not used before) facial over-the-counter or prescription, oral or topical, anti-wrinkle products within 90 days prior to enrolment or planning to begin use of such products at any time during the study.

    NOTE: Continued therapy with some cosmeceuticals (e.g., alpha hydroxyl acids, glycolic acids, retinol, or retinoic acids) is allowed if the regimen was established ≥ 90 days prior to enrolment. The use of sunscreens is also allowed.
15. Known sensitivity to any investigational device or comparator components (see Section 10.1).
16. Previous cosmetic or aesthetic procedures as follows:

    i) All types of previous surgical surgery below the lower orbital rim ii) All types of permanent fillers below the lower orbital rim iii) Previous semi-permanent fillers below the orbital less than 2 years before treatment iv) Previous treatment with HA-based fillers less the 18 months prior to enrolment v) Treatment with photochemotherapy or lasers less than 6 months before enrolment vi) Mechanical, chemical or medical peeling less than 6 months prior to enrolment vii) Treatment with botulinum toxins less than 12 months prior to enrollment viii) Major dental procedures less than 6 months prior to enrolment
17. The presence of abnormal midface function, with inability to effectively puff cheeks, smile broadly, or chew.
18. Pregnant, lactating, or planning to become pregnant at any time during the study.
19. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the investigational device and comparator.
20. History of alcohol or drug abuse or excessive intake of alcohol, as judged by the investigator.
21. Has received any investigational device within 30 days prior to study enrolment or is planning to participate in another investigation during the course of this study.
22. No access to an electronic device (e.g. smartphone, tablet or personal computer) on which to complete eDiaries.
23. Is an employee (or a relative of an employee) of the contract research organization (CRO) responsible for conducting the study, sponsor, or a sponsor representative.
24. The Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the rate of responders determined by the aesthetic improvement of the NLFs according to live on-site evaluator-rated NLF WSRS at 6 months post-treatment between the investigational device and comparator product. | Baseline (pre-treatment) to 6 months post-treatment
  The NLF WSRS is a 5-point scale ranging from 1 (No visible fold; continuous skin line) to 5 (Extremely deep and long folds; detrimental to facial appearance; 2- to 4-mm visible V-shaped fold when stretched). Response is defined as ≥ 1-point improvement on the NLF WSRS for each NLF compared to baseline. Each NLF is to be assessed separately.

SECONDARY OUTCOMES:
Comparison of the rate of responders determined by the aesthetic improvement of the NLFs according to live on-site evaluator-rated NLF WSRS at 1, 3 and 9 months post-treatment between the investigational device and comparator product. | Baseline (pre-treatment) to 1, 3 and 9 months post-treatment
  The NLF WSRS is a 5-point scale ranging from 1 (No visible fold; continuous skin line) to 5 (Extremely deep and long folds; detrimental to facial appearance; 2- to 4-mm visible V-shaped fold when stretched). Response is defined as ≥ 1-point improvement on the NLF WSRS for each NLF compared to baseline. Each NLF is to be assessed separately.
Comparison of the mean change in evaluator-rated NLF WSRS from baseline (pre-treatment) to at 1, 3, 6 and 9 months post-treatment between the investigational device and comparator product. | Baseline (pre-treatment) to 1, 3, 6 and 9 months post-treatment
  The NLF WSRS is a 5-point scale ranging from 1 (No visible fold; continuous skin line) to 5 (Extremely deep and long folds; detrimental to facial appearance; 2- to 4-mm visible V-shaped fold when stretched).
Subject-rated aesthetic improvement in appearance according to GAIS at 1, 3, 6 and 9 months post-treatment. Each NLF is to be assessed separately. | Baseline (pre-treatment) to 1, 3, 6 and 9 months post-treatment
  The 5-grade GAIS assesses the appearance of the NLF compared to pre-treatment on a scale ranging from very much improved to worse.
Evaluating Investigator-rated aesthetic improvement in appearance according to the GAIS at 1, 3, 6 and 9 months post-treatment. Each NLF is to be assessed separately. | Baseline (pre-treatment) to 1, 3, 6 and 9 months post-treatment
  The 5-grade GAIS assesses the appearance of the NLF compared to pre-treatment on a scale ranging from very much improved to worse.
Usability of the device | Baseline - treatment
  Investigator-reported usability of the device. A device usability questionnaire will be completed once by each treating investigator after treatment of his/her last subject.
Subject-reported satisfaction with treatment as assessed by a subject satisfaction questionnaire at 1, 3, 6 and 9 months post-treatment. | 1, 3, 6 and 9 months post-treatment
  Satisfaction will be assessed on a 5-point scale ranging from very satisfied (1) to very dissatisfied (5).
Post-treatment events | Up to 14 days post-treatment
  Incidence, intensity, and duration of pre-defined expected post-treatment events collected using a subject electronic diary (eDiary) for 14 days post treatment.
Adverse Events | Up to 9 months post-treatment
  Frequency, intensity and seriousness of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nilsson, MD, PhD, Principal Investigator — CTC Clinical Trial Consultants AB; Mohammad Alimohammadi, MD, PhD, Principal Investigator — Almo Alo AB
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden